CLINICAL TRIAL: NCT00746954
Title: Buspirone as a Potential Treatment for Recurrent Central Apneas
Brief Title: Buspirone as a Potential Treatment for Recurrent Central Apnea
Acronym: CSA treatment
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Patient recruitment and Funding inadequate to finish trial
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: RESP-006-07F
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Central Apnea; Heart Failure
Keywords: buspirone; acetazolamide
MeSH Terms: conditions — Sleep Apnea, Central; Heart Failure | interventions — Acetazolamide; Buspirone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 BUS to PLA to ACET (Other): Each patient will act as their own control, with comparisons over three nights, each night given buspirone (BUS 20mg), actetazolamide (ACET 250mg), or placebo (PLA) n=3
  Interventions: Drug: Acetazolamide; Drug: Buspirone
- ARM 2 ACET to BUS to PLA (Other): Each patient will act as their own control, with comparisons over three nights, each night given buspirone (BUS 20mg), actetazolamide (ACET 250mg), or placebo (PLA) n=3
  Interventions: Drug: Acetazolamide; Drug: Buspirone
- ARM 3 PLA to ACET to BUS (Other): Each patient will act as their own control, with comparisons over three nights, each night given buspirone (BUS 20mg), actetazolamide (ACET 250mg), or placebo (PLA) n=2
  Interventions: Drug: Acetazolamide; Drug: Buspirone

INTERVENTIONS:
Drug: Acetazolamide — Cabonic Anhydrase inhibitor
Drug: Buspirone — Agonist of a 5-HT1a receptor with some D2 agonist properties.

SUMMARY:
The purpose of this study is to determine whether buspirone compared to acetazolamide and to placebo will reduce the number and/or severity of breathing pauses during sleep that occur in some patients with Heart Failure.

DETAILED DESCRIPTION:
The hypothesis is that buspirone is a safe, effective drug to reduce the occurrence of recurrent central apnea and irregular breathing found in the setting of heart failure. A secondary hypothesis is that its effect will be similar to that or acetazolamide. Study Design: A one-dose double-blind crossover study of buspirone vs. placebo vs. acetazolamide will be performed to determine if active drug alters the number and/or severity of recurrent central apneas and hypopneas (AHI) in patients with heart failure. AHI is the primary outcome variable. In the initial phase of this study, we will recruit 18-20 patients to obtain ~15 complete studies, using the assumption of a ~20% drop-out, to reach a pre-set significance level of a 30% reduction in AHI in the drug groups with a power of 0.90 and a p=0.05 by post-hoc testing. Power estimates were calculated using the means and SDs derived from the population reported the study of acetazolamide by Javaheri et al (2006). A 30% reduction in AHI would be meaningful. A 15% dropout rate was present in the study by Javaheri et al (2006), but as our study is a three-way comparison, we chose a slightly higher rate. The reasons stated in these articles for a drop out included: viral illness, GI upset (on placebo or on theophyllin), tired of the sleep studies, and desire to terminate without cause. Statistical Analyses. Analysis of variance for repeated measures using Sidak's correction will be used to compare placebo, buspirone, and acetazolamide studies. For variables that are not normally distributed, Dunn's nonparametric test for multiple comparisons will be used. p > 0.05 will be considered significant. Mean values and SDs will be reported. This single dose, one night study is called Buspirone as a Potential Treatment for Recurrent Sleep Apnea I.

The randomization will be in a block design, and the analysis will take into account the blocked design. We will recruit 30 patients to obtain ~27 complete studies, using the assumption of a ~25% drop-out, to reach a pre-set significance level of a 50% reduction in AHI in the drug groups with a power of 0.90 and a p=0.05 by post-hoc testing (see Table C below). Power estimates were calculated using the means and SDs derived from the population reported the study of a one week trial of acetazolamide by Javaheri, values similar to those in the drug trial for theophyllin. Our reasoning is that a 50% reduction in AHI would be most meaningful. Our drop-out rate in the one-night study is estimated at ~25%.

Exclusion criteria of use of selective serotonin reuptake inhibitors (SSRIs) or antidepressants, while necessary because one of the drugs was buspirone, were too stringent for completion of this study in the VA setting. Of ~1000 patient charts screens, 8 were eventually entered into the trial, so that power criteria were not met. Records are being utilized to probe for hidden features in the PSG for use in future drug trials.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent,
* Ambulatory and in stable condition for the past 4 months,
* A diagnosis of heart failure with left ventricular systolic dysfunction as evidenced by an ejection fraction <35%,
* NYHA class II or III clinical status, and
* Diagnosis of dilated cardiomyopathy or ischemic cardiomyopathy.

Exclusion Criteria:

* Unstable angina, unstable heart failure, acute pulmonary edema, congenital heart disease
* History of unstable and/or advanced hepatic disease
* History of renal failure, CrCL < 30
* Current use of an SSRI, or use within one month of testing
* Intrinsic pulmonary diseases: ILD and/or COPD (FEV1/FVC < 65%)
* Kyphoscoliosis or neuromuscular disease
* Suboptimally treated hypothyroidism
* Use of narcotics or benzodiazepines
* Use of theophylline or pseudoephedrine
* Use the following medications:

  * MAO inhibitors
  * diazepam
  * haloperidol
  * nefazodone
  * trazodone
  * erythromycin
  * grapefruit juice
  * itraconazole
  * rifampin
  * ketoconazole
  * ritonavir,
  * cimetidine
* Known allergy to buspirone or acetazolamide

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-09; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kingman P. Strohl, MD, Principal Investigator — VA Medical Center-Cleveland
Locations (1):
- VA Medical Center, Cleveland, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the VA.
Pre-assignment Details: The HF population has psychiatric co-morbidity and often is empirically treated with antidepressants.
  We screened >1000 records but enrolled and completed 8 patients, before running out of resources.
Groups:
- Arm 1 Control to ACET to BUS: Each patient will act as their own control, with comparisons over three nights, this is placebo
- Arm 2 Acet to Placebo to Bus: Each patient will act as their own control, with comparisons over three nights, each night given actetazolamide (Acet 250mg), or placebo or buspirone (Bus 20mg),
- Arm 3 BUS to ACET to PLA: Each patient will act as their own control, with comparisons over three nights, each night given buspirone (20mg), actetazolamide (250mg), or placebo
Period: Overall Study
Arm/Group | Arm 1 Control to ACET to BUS | Arm 2 Acet to Placebo to Bus | Arm 3 BUS to ACET to PLA
Started | 3 | 3 | 2
Completed | 3 | 3 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Each patient will act as their own control, with comparisons over three nights, each night given buspirone (20mg), actetazolamide (250mg), or placebo
Arm/Group | Arm 1
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Apnea-hypopnea Index (Number of Central and Mixed Apneas/Hour of Sleep)
Time Frame: Overnight polysomnogram over 3 separate nights
Population: Comparisons among Drugs (not Arms)
Measure: Mean (Standard Deviation); unit: APNEA-HYPOPNEA/HR by drug or placebo
Groups:
- BUSPIRONE: Each patient will act as their own control, with comparisons over three nights, each night given buspirone (20mg), actetazolamide (250mg), or placebo
- ACETAZOLAMIDE; PLACEBO: Each patient will act as their own control, with comparisons over three nights
Arm/Group | BUSPIRONE | ACETAZOLAMIDE | PLACEBO
Number analyzed (Participants) | 8 | 8 | 8
APNEA-HYPOPNEA/HR by drug or placebo | 32.5 (5) | 31.2 (4.9) | 35.7 (8)
Statistical Analysis 1: Comparison: BUSPIRONE vs ACETAZOLAMIDE vs PLACEBO; Comparisons among groups; Test type: Superiority or Other; p = 0.45, ANOVA

ADVERSE EVENTS:
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
VA population turned out to have a high number of heart failure patients who had psychiatric co-morbidity or were empirically treated with antidepressants, precluding participation.

There were not enrolled enough participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes